CLINICAL TRIAL: NCT06246279
Title: The Effect of the Education Program Prepared in Line With Transition Theory on Adaptation to Adolescence and Disease Management in Adolescents With Type 1 Diabetes: Randomized Controlled Study
Brief Title: Disease Management in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ceren Calik, Master of Science, specialist nurse, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AdolescentswithType1Diabete
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: type1diabetes; Adolescent Behavior; Self Efficacy
Keywords: Type 1 Diabetes; Transition Theory; Diabetes Management; Pediatric Nurse; Randomized Controlled Trial
MeSH Terms: conditions — Adolescent Behavior; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In addition to the institution's routine T1DM training, the "Adjustment to Adolescence and Transition to Type 1 Diabetes Education Program" prepared in line with Meleis's Transition Theory was applied to adolescents online via the Microsoft Teams Program.
  Interventions: Behavioral: Adaptation to Adolescence and Type 1 Diabetes Management Training Program
- Control group (No Intervention): The institution's routinely planned diabetes education was given by the pediatric diabetes education nurse.

INTERVENTIONS:
Behavioral: Adaptation to Adolescence and Type 1 Diabetes Management Training Program — The content of the Training Program was created by researchers based on Transition Theory, in line with high-level research results and international guides. Then, the necessary arrangements were made by taking the opinions of 10 experts (child health and disease nursing faculty member, child and adolescent mental health specialist, child endocrinologist, child development specialist, nutrition and dietetics specialist, sports training specialist). The content was finalized in line with the comments received.
  Arms: Experimental group

SUMMARY:
Adolescence period; It is a transition period of rapid growth, development and maturation in biochemical, physical, social and spiritual terms, which lasts from the beginning of puberty to young adulthood. Adolescence is a predictable developmental transition period for the individual. They also encounter unpredictable situations (such as childhood illnesses). One of these conditions is Type 1 Diabetes Mellitus, which is the most common metabolic endocrine system disease in adolescents. Type 1 diabetes is an important health/disease transition in the life of a child and adolescent. Therefore, this study aimed to determine the effect of the "Adaptation to Adolescence and Type 1 Diabetes Management Training Programme", prepared in line with Meleis's Transition Theory, on the adolescent's developmental transition adaptation, self-efficacy for diabetes management and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with type 1 diabetes in the last 6 months
* HbA1c level >7.5

Exclusion Criteria:

* presence of a diagnosis of intellectual disability, autism spectrum disorder and psychotic disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Reynolds Adjustment Screening Inventory for Adolescents | This scale was administered three times at beginning, 3rd and 6th months.
  Reynolds Adjustment Screening Inventory has four subscales. These; emotional distress (10 items), antisocial behavior (8 items), positive self (6 items related to self-confidence and socialization) and anger control problems (8 items). The Cronbach alpha value of the scale is stated as 0.91. The lowest score of the scale is 32 and the highest score is 165.

SECONDARY OUTCOMES:
Diabetes Management Self-Efficacy Scale in Adolescents with Type 1 Diabetes | This scale was administered three times at beginning, 3rd and 6th months.
  The scale is used to determine the educational needs of adolescents or to evaluate the effectiveness of diabetes education programs. The scale consists of 26 items ranging from 1 (completely agree) to 5 (strongly disagree). The lowest total score that can be obtained from the scale is 26 and the highest is 130. A higher score indicates less self-efficacy. The Cronbach's alpha coefficient of the scale was found to be 0.85.
Glycemic Control - Hemoglobin A1C | This scale was administered three times at beginning, 3rd and 6th months.
  Glycemic control was assessed by HbA1C level. In Type 1 Diabetes, Hb A1C level is one of the basic control parameters checked in the clinic in adolescents. It is repeated routinely every 3 months when the child comes to the outpatient clinic for control for Type 1 Diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Calik, Principal Investigator — Akdeniz Univercity
Locations (1):
- Akdeniz Univercity, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No